CLINICAL TRIAL: NCT02787785
Title: Multicenter Automatic Defibrillator Implantation Trial With Subcutaneous Implantable Cardioverter Defibrillator (MADIT S-ICD)
Brief Title: Multicenter Automatic Defibrillator Implantation Trial With Subcutaneous Implantable Cardioverter Defibrillator
Acronym: MADIT S-ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MADIT S-ICD (C1834)
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Tachycardia; Diabetes Mellitus; Cardiovascular Disease
Keywords: Subcutaneous; Implantable Cardioverter Defibrillator; MADIT; Diabetes; Myocardial Infarction
MeSH Terms: conditions — Tachycardia; Diabetes Mellitus; Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional Medical Therapy (No Intervention): This arm of the trial continues with their current conventional medical therapy.
- Subcutaneous Implantable Cardioverter Defibrillator (Active Comparator): This arm of the trial receives a subcutaneous implantable defibrillator.
  Interventions: Device: Subcutaneous Implantable Cardioverter Defibrillator

INTERVENTIONS:
Device: Subcutaneous Implantable Cardioverter Defibrillator — The S-ICD is an entirely subcutaneous implantable cardioverter defibrillator.
  Arms: Subcutaneous Implantable Cardioverter Defibrillator

SUMMARY:
The MADIT S-ICD trial was designed to evaluate if subjects with a prior myocardial infarction, diabetes mellitus and a relatively preserved ejection fraction of 36-50% will have a survival benefit from receiving a subcutaneous implantable cardioverter defibrillator (S-ICD) when compared to those receiving conventional medical therapy. The trial enrollment was stopped in 2018 due to lower than expected enrollment, all subjects enrolled at that time were followed for approximately 5 years.

DETAILED DESCRIPTION:
In this study, subjects were randomized to receive a subcutaneous implantable cardioverter defibrillator or Conventional Medical Therapy (CMT). Randomization was stratified by enrolling site, in a 2:1 (S-ICD:CMT) scheme. Length of follow-up for each subject was dependent on the date of entry into the study, since all subjects were followed to a common study termination date.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years on date of consent
* Diabetes mellitus treated with oral hypoglycemic agents, non-insulin injectable and/or insulin for the past 3 calendar months or longer prior to consent date
* LV ejection fraction (LVEF) of 36-50% documented by imaging (preferably by MRI or echocardiographic methods), within 12 calendar months before consent date and at least 3 calendar months after most recent Myocardial Infarction (MI), percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG).
* One or more clinically documented, enzyme-positive myocardial infarctions, more than 3 calendar months prior to consent date*. (If enzyme information and clinical documentation is not available, there must be a clear evidence of prior silent myocardial infarction identified as either new pathologic Q waves on ECG or imaging documentation of an infarcted area (left ventricular angiography/ nuclear scan/ MRI) Note: MI qualification based on the Universal Definition of MI)
* Qualifying 12-lead ECG within 6 calendar months before consent date and at least 3 calendar months after most recent MI, PCI or CABG. (The qualifying ECG* can be sinus rhythm or atrial fibrillation (patients with persistent or permanent atrial fibrillation should have a controlled ventricular response <100 bpm on consent date) *QRS duration on the qualifying ECG >90 msec)
* Passing S-ICD Screening ECG performed per applicable user's manual on or after the consent date that identifies one or more qualifying S-ICD sensing vectors

Exclusion Criteria:

* Ejection fraction >50% or <36% within 12 calendar months prior to consent date and at least 3 calendar months after the most recent MI, PCI or CABG
* Existing guideline based indication for an implantable cardioverter defibrillator (ICD), pacemaker, cardiac resynchronization therapy device (CRT), or cardiac resynchronization therapy device with defibrillator (CRT-D) therapy
* Existing or previously implanted ICD, CRT, CRT-D, or pacemaker device system
* Active infection at the time of consent
* Contraindication for S-ICD implantation according to the S-ICD pulse generator (PG) User's Manual
* Hemodialysis and/or peritoneal dialysis at the time of enrollment
* New York Heart Association Class IV in the past 3 calendar months prior to or at the time of consent date
* Coronary artery bypass graft surgery or percutaneous coronary intervention (balloon and/or stent angioplasty) within 3 calendar months prior to the consent date
* Enzyme-positive myocardial infarction or silent myocardial infarction diagnosed within 3 calendar months prior to the consent date
* Unstable angina with need for outpatient treatment or hospitalization (change/addition of anti-anginal medication and/or coronary revascularization), within 3 calendar months prior to the consent date
* Angiographic evidence of coronary disease in a patient that is a candidate for coronary revascularization and is likely to undergo CABG or PCI in the next 3 calendar months
* High risk for arterial embolism (e.g. presence of mobile left ventricular thrombus)
* Hemodynamically significant congenital heart disease, aortic valvular heart disease, or amyloid heart disease
* Baseline body mass index > 45 kg/m2
* On a heart transplant list or likely to undergo heart transplant within one calendar year
* Presence of any other disease, other than the subject's cardiac disease, that in the opinion of the investigator is likely to significantly reduce the patient's likelihood of survival for the duration of the trial (e.g. cancer, liver failure).
* Unwillingness or inability to cooperate with the protocol
* Resides at such a distance from the enrolling site so travel to follow-up visits would be unusually difficult
* Reversible causes of heart disease (e.g. viral myocarditis or tachycardia induced cardiomyopathy)
* Participation in other clinical trials (observational registries are allowed with approval from the CDC)
* Does not anticipate residing in the vicinity of the enrolling site for the duration of the trial
* Unwillingness to sign the consent for participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD, MSc, PhD, Principal Investigator — University of Rochester Heart Research Follow-up Program
Locations (49):
- United States (36):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Glendale Adventist Medical Center, Glendale, California
  - University of Southern California, Los Angeles, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - Alta Bates Summit Hospital, Oakland, California
  - Huntington Hospital, Pasadena, California
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Cardiovascular Associates of Delaware Valley, Haddon Heights, New Jersey
  - Northwell Health, Manhasset, New York
  - Strong Memorial / University of Rochester Medical Center, Rochester, New York
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Ohio State Wexner Medical Center, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Promedica Toledo Hospital, Toledo, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - University of Pittsburgh Medical Center - Presbyterian, Pittsburgh, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - University of Texas, Houston, Houston, Texas
  - Sentara Norfolk General, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
- Germany (3):
  - Medizinische Hochschule Hannover, Hannover, Lower Saxony
  - Unfallkrankenhaus Berlin, Berlin
  - Universitaetsklinik Eppendorf, Hamburg
- Israel (3):
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Azienda Ospedaliera Ospedale Niguarda CA Granda, Milan, Niguarda
  - Azienda Ospedaliera Universitaria, Verona
- Netherlands (2):
  - UMC Utrecht, Utrecht, CX
  - Academisch Medisch Centrum, Amsterdam, North Holland
- Spain (2):
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - University of Navarra, Department of Cardiology, Pamplona, Navarre
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kutyifa V, Beck C, Brown MW, Cannom D, Daubert J, Estes M, Greenberg H, Goldenberg I, Hammes S, Huang D, Klein H, Knops R, Kosiborod M, Poole J, Schuger C, Singh JP, Solomon S, Wilber D, Zareba W, Moss AJ; MADIT S-ICD Executive Committee. Multicenter Automatic Defibrillator Implantation Trial-Subcutaneous Implantable Cardioverter Defibrillator (MADIT S-ICD): Design and clinical protocol. Am Heart J. 2017 Jul;189:158-166. doi: 10.1016/j.ahj.2017.04.014. Epub 2017 May 4. PMID 28625372

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Medical Therapy | Subcutaneous Implantable Cardioverter Defibrillator
Started | 11 | 29
Completed | 7 | 19
Not Completed | 4 | 10
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Conventional Medical Therapy: This arm of the trial continued with current conventional medical therapy.
- Subcutaneous Implantable Cardioverter Defibrillator: This arm of the trial received a subcutaneous implantable defibrillator.
  Subcutaneous Implantable Cardioverter Defibrillator: The S-ICD is an entirely subcutaneous implantable cardioverter defibrillator.
- Total: Total of all reporting groups
Arm/Group | Conventional Medical Therapy | Subcutaneous Implantable Cardioverter Defibrillator | Total
Number analyzed (Participants) | 11 | 29 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (5.0) | 71.1 (4.7) | 70.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 11 | 26 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 8 | 24 | 32
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 27 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 22 | 28
  Israel | 2 | 3 | 5
  Germany | 2 | 1 | 3
  Spain | 1 | 3 | 4
New York Heart Association Class (NYHA) [Count of Participants; unit: Participants] — Subject NYHA Class was collected from the participant's medical record. The American Heart Association, definitions are: Class I is no limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath. Class II is Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain. Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  Participants
    NYHA Class I | 2 | 6 | 8
    NYHA Class II | 8 | 21 | 29
    NYHA Class III | 1 | 2 | 3
History of Atrial Fibrillation [Count of Participants; unit: Participants] | 2 | 8 | 10
History of Ventricular Arrhythmias [Count of Participants; unit: Participants] | 1 | 6 | 7
Prior CHF Hospitalization [Count of Participants; unit: Participants] | 3 | 7 | 10
Prior Coronary Artery Bypass Graft [Count of Participants; unit: Participants] | 6 | 10 | 16
Prior Percutaneous Coronary Intervention [Count of Participants; unit: Participants] | 9 | 19 | 28
Hypertension [Count of Participants; unit: Participants] | 11 | 24 | 35

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Mortality
Description: The original study design was event driven with the end date expected to be based on crossing the statistical boundary. The trial enrollment was stopped in 2018 due to lower than expected enrollment, all subjects enrolled at that time were followed for approximately 5 years. The outcomes will be analyzed but are no longer statistically powered for conclusions.
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Medical Therapy | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 11 | 29
Participants | 3 | 4
Statistical Analysis 1: Comparison: Conventional Medical Therapy vs Subcutaneous Implantable Cardioverter Defibrillator; Test type: Superiority; p = 0.354, Regression, Cox; Cox Proportional Hazard = 0.49, 95% CI 2-sided [0.11 to 2.20]

2. Secondary Outcome: All-Cause Mortality in Various Subgroups
Description: as for outcome 1
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Population: Multiple sub-groups had insufficient number of patients and/or events for analyses. Therefore, interaction analyses are not provided. The secondary endpoint is limited to the following subgroups: gender, race, ethnicity, age dichotomized at 70 years, left ventricular ejection fraction (LVEF) dichotomized at 40%, duration of diabetes, presence versus absence of insulin therapy, HbA1c dichotomized at 8%, and QRS duration > 120 milliseconds (ms).
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Medical Therapy | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 11 | 29
Participants
  Men: number analyzed (Participants) | 11 | 26
  Men | 3 | 2
  Women: number analyzed (Participants) | 0 | 3
  Women | 0 | 2
  Race - White: number analyzed (Participants) | 9 | 27
  Race - White | 3 | 3
  Race - African American: number analyzed (Participants) | 0 | 2
  Race - African American | 0 | 1
  Ethnicity - Non-Hispanic: number analyzed (Participants) | 8 | 24
  Ethnicity - Non-Hispanic | 3 | 3
  Ethnicity - Hispanic: number analyzed (Participants) | 2 | 5
  Ethnicity - Hispanic | 0 | 1
  Age </= 70 years: number analyzed (Participants) | 8 | 16
  Age </= 70 years | 2 | 2
  Age > 70 years: number analyzed (Participants) | 3 | 13
  Age > 70 years | 1 | 2
  LVEF </= 40%: number analyzed (Participants) | 3 | 12
  LVEF </= 40% | 1 | 3
  LVEF > 40%: number analyzed (Participants) | 8 | 17
  LVEF > 40% | 2 | 1
  Insulin Therapy: number analyzed (Participants) | 7 | 15
  Insulin Therapy | 2 | 3
  No Insulin Therapy: number analyzed (Participants) | 4 | 14
  No Insulin Therapy | 1 | 1
  Diabetes duration</= 2 years: number analyzed (Participants) | 4 | 14
  Diabetes duration</= 2 years | 1 | 1
  Diabetes duration > 2 years: number analyzed (Participants) | 4 | 10
  Diabetes duration > 2 years | 1 | 3
  HbA1c </= 8 %: number analyzed (Participants) | 7 | 20
  HbA1c </= 8 % | 2 | 4
  HbA1c > 8 %: number analyzed (Participants) | 2 | 2
  HbA1c > 8 % | 0 | 0
  QRS </= 120ms: number analyzed (Participants) | 8 | 23
  QRS </= 120ms | 2 | 3
  QRS > 120ms: number analyzed (Participants) | 3 | 6
  QRS > 120ms | 1 | 1

3. Secondary Outcome: Sudden Death
Description: as for outcome 1
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Medical Therapy | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 11 | 29
Participants | 1 | 1
Statistical Analysis 1: Comparison: Conventional Medical Therapy vs Subcutaneous Implantable Cardioverter Defibrillator; Test type: Superiority; p = 0.479, Regression, Cox; Cox Proportional Hazard = 0.37, 95% CI 2-sided [0.02 to 5.88]

4. Other Pre Specified Outcome: S-ICD Inappropriate Shock Frequency
Description: Pre-specific tertiary statistical analyses will be descriptive and exploratory. This describes the number of inappropriate shocks received in the study .
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Measure: Number; unit: inappropriate shocks
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 29
inappropriate shocks | 5

5. Other Pre Specified Outcome: S-ICD Inappropriate Shock Outcomes
Description: Pre-specific tertiary statistical analyses will be descriptive and exploratory. This describes the percent of participants that received an inappropriate shock.
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 29
Participants | 4

6. Other Pre Specified Outcome: S-ICD Treated Ventricular Arrhythmia Frequency
Description: Pre-specific tertiary statistical analyses will be descriptive and exploratory. This describes the number of appropriate shocks received during the study.
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Measure: Number; unit: appropriate device shocks
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 29
appropriate device shocks | 5

7. Other Pre Specified Outcome: S-ICD Treated Ventricular Arrhythmia Outcomes
Description: Pre-specific tertiary statistical analyses will be descriptive and exploratory. This describes the number of participants that received an appropriate shock.
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 29
Participants | 3

8. Other Pre Specified Outcome: S-ICD Device Complications
Description: Pre-specific tertiary statistical analyses will be descriptive and exploratory.
Time Frame: Outcome measured timeframe includes all available follow-up. Median 61 (4, 71) months.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Subcutaneous Implantable Cardioverter Defibrillator
Number analyzed (Participants) | 29
percentage of patients | 21 [10.1 to 41.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization through to a common end date with the minimum amount of follow-up time being 5-years. The Median follow-up time for participants was 61 months.
Arm/Group | Conventional Medical Therapy | Subcutaneous Implantable Cardioverter Defibrillator
All-Cause Mortality (participants affected / at risk) | 3/11 | 4/29
Serious Adverse Events (participants affected / at risk) | 8/11 | 20/29
Other Adverse Events (participants affected / at risk) | 4/11 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Medical Therapy (N=11) | Subcutaneous Implantable Cardioverter Defibrillator (N=29)
Inappropriate tachy therapy (Product Issues) | 0 (0) | 1 (1)
Incisional/Superficial infections (</= 30 days post implant without explant) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hematoma - Device pocket (> 30 days post implant) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device System Discomfort (> 30 days post implant) (Product Issues) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea - Heart Failure (Cardiac disorders) | 1 (1) | 2 (2)
Pulmonary Edema - Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Heart Failure Symptoms, unspecified (Cardiac disorders) | 1 (1) | 2 (2)
Multiple Heart Failure Symptoms (Cardiac disorders) | 1 (1) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 2 (3) | 5 (5)
Peripheral Vascular Disease (Vascular disorders) | 2 (4) | 1 (1)
Pseudoaneurysm without hematoma (Vascular disorders) | 1 (1) | 0 (0)
Aortic Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 2 (2)
Chest Pain - Ischemic (Cardiac disorders) | 1 (1) | 3 (4)
Chest Pain- Other (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue/Weakness (General disorders) | 0 (0) | 1 (1)
Subject Condition - Cardiovascular (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (CVA) - unspecified (Vascular disorders) | 0 (0) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death, unknown cause (Cardiac disorders) | 0 (0) | 1 (1)
Systemic Infection (Infections and infestations) | 0 (0) | 5 (5)
Fever and or virus (General disorders) | 0 (0) | 2 (2)
Physical Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Localized Infection (Infections and infestations) | 1 (1) | 2 (2)
Hematological (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neurological (Nervous system disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (8)
Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal (Renal and urinary disorders) | 0 (0) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Endocrine (Endocrine disorders) | 0 (0) | 1 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Medical Therapy (N=11) | Subcutaneous Implantable Cardioverter Defibrillator (N=29)
Inappropriate tachy therapy, noise (Product Issues) | 0 (0) | 3 (3)
Inappropriate therapy - SVT discrimination error - System (Product Issues) | 0 (0) | 2 (3)
Inadvertent Arrhythmia - Procedure (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Chest Pain - other (General disorders) | 2 (2) | 1 (2)
Physican Trauma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Neurological (Nervous system disorders) | 2 (2) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The primary limitation for MADIT S-ICD was the enrollment stop. The study intended to enroll 1800 subjects; however enrollment was stopped due to slow patient recruitment. The 40 subjects enrolled prior to stopping were followed for a minimum of 5 years for safety. Statistics performed and outcomes included are observational and no longer powered for assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT02787785/Prot_SAP_000.pdf